CLINICAL TRIAL: NCT05667766
Title: Minimising Adverse Drug Reactions and Verifying Economic Legitimacy - Pharmacogenomics Implementation in Children (MARVEL-PIC)
Brief Title: Minimising Adverse Drug Reactions and Verifying Economic Legitimacy in Children (MARVEL-PIC)
Acronym: MARVEL-PIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 89083
Record Dates: First submitted 2022-12-19; First posted 2022-12-29 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Neoplasms; Bone Marrow Transplantation
Keywords: cancer; paediatric; pharmacogenomic
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Other): Standard of Care prescribing for period of 12 months. Participants will receive pharmacogenomic test results according to the current standard of care. The participants will be followed up for a minimum of 12 weeks, with maximal time-period being 12 months depending on time of enrolment.
  Interventions: Diagnostic Test: Release of Extended Pharmacogenomics Report at Week 13
- Experimental Arm (Experimental): Extended Pharmacogenomic prescribing for a period of 12 months. Participants will receive pharmacogenomic testing across a range of clinically relevant variants, to guide the dose and drug selection of 27 drugs commonly used in supportive care. The participants will be followed up for a minimum of 12 weeks, with maximal time-period being 12 months depending on time of enrolment.
  Interventions: Diagnostic Test: Release of Extended Pharmacogenomics Report at Week 1; Diagnostic Test: Release of Extended Pharmacogenomics Report at Week 13

INTERVENTIONS:
Diagnostic Test: Release of Extended Pharmacogenomics Report at Week 1 — Whole genome sequencing with reporting on current standard of care (SoC) pharmacogenomic variants (TPMT, NUD15) where applicable (i.e, for patients with diagnosis of acute lymphoblastic leukaemia) by Week 1. Whole genome sequencing on a broader number of actionable variants as per international guidelines for cancer supportive care (identical to study arm) will be reported on at Week 13.
  Arms: Experimental Arm
Diagnostic Test: Release of Extended Pharmacogenomics Report at Week 13 — Whole genome sequencing with reporting on current standard of care (SoC) pharmacogenomic variants (TPMT, NUD15) where applicable (i.e, for patients with diagnosis of acute lymphoblastic leukaemia) and reporting of a broader number of actionable pharmacogenomic variants as per international guidelines for cancer supportive care reported on by Week 1.

SUMMARY:
A prospective, open, randomised implementation study in paediatric cancer patients. The study aims to determine whether a personalised approach will result in an overall reduction in clinically relevant adverse drug reactions (ADRs) and to evaluate the economic and quality of life impacts. Participants will be randomised to receive personalised guided prescribing of supportive care therapy (study arm) or standard of care (control arm) for a period of 12 weeks. The follow up period includes prospective patient reporting of symptoms and quality of life through electronically delivered surveys, for a maximum of 12 months.

DETAILED DESCRIPTION:
One of the main areas of precision medicine that is easily implementable is pharmacogenomic testing. Germline testing of genes predisposing to drug toxicity or inefficacy can inform drug selection and dosing. This steers away from the historical 'trial and error' approach, avoids unnecessary adverse drug reactions (ADRs) and can potentially impact on health economic savings, through reduction in readmissions and admissions with ADRs.

This study will be a prospective, open, randomised implementation study in paediatric and adolescent patients with a new diagnosis of cancer or who are proceeding to first haematopoietic stem cell transplantation (HSCT). The current standard of care for paediatrics in Australia involves pharmacogenomic testing for TPMT and NUD15, for patients with acute lymphoblastic leukaemia. Participants of the study will receive pharmacogenomic testing across a range of clinically relevant variants. Participants will be randomised to either the control arm or the study arm. Test results for participants in the study arm will be used to guide the dose and drug selection of 27 drugs commonly used in supportive care. The pharmacogenomic test results will be released to the study arm at week 4 and to the control arm at week 13, after the 12 week intervention period.

To determine whether pre-emptive pharmacogenomic testing does reduce clinically relevant adverse drug reactions, the Paediatric Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (Ped-PRO-CTCAE) survey will be delivered at 3 time points within a 12 week period. This survey is a patient reported outcome measurement tool developed to evaluate symptomatic toxicity in participants receiving cancer therapy. After survey completion, semi-structured interviews will be conducted by an academic pharmacist with the aim of generating a CTCAE grade of severity for each of the symptoms defined in the Ped-PRO-CTCAE and assessing the causality of an adverse drug reaction using the Liverpool Adverse Drug Reaction Causality Assessment Tool (Liverpool ADR-CAT). These mechanisms will support the assessment of both severity and causality of any adverse drug reactions.

To evaluate the economic and Quality of Life impacts (QoL), participants will also complete The Child Health Utility 9D (CHU9D) QoL surveys specific to children and young adults at 3 timepoints over the 12-month period and consent to a Health Economics Analysis. This includes collection of Medicare Benefits Schedule (MBS)/ Pharmaceutical Benefits Scheme (PBS) data from Services Australia and Victorian Data Linkage Group to compare the costs of management of both the control and study arm.

Data from the study will be securely stored on the REDCap database. Patients will be allocated a unique patient identifier prior to their de-identified data being added to the database.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years
* New cancer diagnosis or patient receiving HSCT or patient has a relapsed cancer diagnosis and is starting treatment after more than 6 months without.
* Starting treatment with a chemotherapeutic agent that is not single agent oral targeted therapy.
* Must also be taking a medication for which there is an established CPIC guideline available.
* Parent or patient is able and willing to give consent for patient to take part and be followed up for at least 12 weeks.
* Patient is amenable to venepuncture and blood draw (5mL ideally with an absolute minimum requirement of 2.5 mL) or has Whole Genome Sequencing available (WGS).
* Patient and/or parent is able and willing to sign an informed consent form.
* Patient and/or parent is able to complete Ped-PRO-CTCAE survey in English, Italian or Chinese.
* Study enrolment limit has not been reached.

Exclusion Criteria:

* Age > 18 years.
* Patient has a life expectancy estimated to be less than three months by the treating clinical team.
* Duration of the drug of inclusion total treatment length is planned to be less than one week.
* Patient and/or parent is unable to consent to the study.
* Patient and/or parent is unwilling to take part in the study.
* Patient and/or parent is able unable to complete Ped-PRO-CTCAE survey in English, Italian or Chinese.
* Patient has existing impaired hepatic or renal function for which a lower dose or alternate drug selection are already part of current routine care.
* Patient has a glomerular filtration rate of less than 15 mL/min per 1.73m2.
* Patient has advanced liver failure.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 880 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Reduction in the number of adverse drug reactions (ADRs) | 12 weeks
  The primary outcome is a reduction in adverse drug reactions among patients with actionable pharmacogenomic variants. An adverse drug reaction will be considered as any CTCAE grade 2 and above for non-haematological toxicities or CTCAE grade 3 and above for haematological toxicities. CTCAE grades are defined as 1,2,3,4 or 5, with 5 indicating the most severe.

SECONDARY OUTCOMES:
Occurrence of at least one ADR which contributes to primary endpoint | 12 weeks
  An adverse drug reaction will be considered as any CTCAE grade 2 and above for non-haematological toxicities or CTCAE grade 3 and above for haematological toxicities. This includes an ADR which was caused either by the index drug of inclusion or any subsequent drug. CTCAE grades are defined as 1,2,3,4 or 5, with 5 indicated the most severe.
Occurrence of at least one causal, clinically relevant, drug-genotype specific ADR, attributable to the index drug. | 12 weeks
  The Liverpool ADR CAT is an assessment tool produced to attribute causality to specific drugs for the grading of ADR symptomatic toxicity. Possible grading of ADRs include either definite, probable or possible.
Number of self-reported ADRs | 12 weeks
  The Ped-PRO-CTCAE survey is an electronic patient reported outcome measurement survey developed to evaluate symptomatic toxicity in patients who are receiving cancer therapy. Symptoms are evaluated for attributes of frequency, severity, interference, amount, presence or absence. Each symptomatic adverse event (AE) is assessed by 1-3 attributes that can be linked back to a CTCAE grade. The number of self-reported ADRs are measured independent of severity or drug-gene association but caused by one of the chemotherapeutic /targeted agents.
Number of serious self-reported ADRs | 12 weeks
  The Ped-PRO-CTCAE survey is an electronic patient reported outcome measurement survey developed to evaluate symptomatic toxicity in patients who are receiving cancer therapy. Symptoms are evaluated for attributes of frequency, severity, interference, amount, presence or absence. Each symptomatic adverse event (AE) is assessed by 1-3 attributes that can be linked back to a CTCAE grade. The number of self-reported ADRs are measured independent of severity or drug-gene association but caused by one of the chemotherapeutic /targeted agents. An ADR will be classified as serious if that event led to death, serious deterioration in health, or fetal distress.
Number of dose adjustments | 12 weeks
  Number of dose adjustments made to drug-gene associated therapy during the entire study follow up by review of the participants electronic medical record and medication reconciliation.
Incidence of drug cessation due to ADR | 12 months
  Incidence of drug cessation due to ADR during the entire study follow up. Relates to inclusion criteria drug by review of the participants electronic medical record and medication reconciliation.
Incidence of drug cessation due to lack of efficacy | 12 months
  Incidence of drug cessation due to lack of efficacy by review of the participants electronic medical record and medication reconciliation.
Therapeutic drug monitoring | 12 months
  Therapeutic drug monitoring (routine drug levels) performed during entire study follow up period by review of the participants electronic medical record and medication reconciliation.
Physician and Pharmacist adherence to the CPIC guidelines | 12 months
  After discussion and consensus of a pharmacogenetic variant. A clinical report will be generated with the results and therapeutic recommendations according to Clinical Pharmacogenetics Implementation Consortium (CPIC) guidelines. Adherence to recommendations will be reported with reasoning, during the 12 week period.
Health care expenditure related to adverse events using MBS/PBS data | 12 months
  Data will be collected on the costs of management comparing the standard of care arm versus the study arm. The actual costs assigned to each inpatient or outpatient episode will be collected. This information is readily accessible through Services Australia and The Department of Health via The Centre for Victorian Data Linkage (CVDL).
Change in quality of life outcomes using CHU9D | Baseline, Week 12, 12 months
  The University of Sheffield CHU9D Quality of Life Survey will be used to monitor changes in patient QoL. The CHU9D consists of a descriptive system and set of preference weights, for 9 questions that assess participants daily functioning across the following domains: worry, sadness, pain, tiredness, annoyance, school, sleep, daily routine and activities. The tool allows for calculation of quality adjusted life years for use in cost utility analysis

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Rachel Conyers, Principal Investigator — The Royal Children's Hospital/Murdoch Children's Research Institute
Locations (4):
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Women's and Children's Hospital, North Adelaide, South Australia
  - The Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Washington

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the study will be available from 6 months after publication of the primary outcome. Only de-identified data will published. The study protocol, analysis plan and consent forms will also be available. The data may be obtained from the Murdoch Children's Research Institute by emailing MCTC@mcri.edu.au.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified data set collected for the analysis of the trial will be available from six months after publication of the primary outcome. The study protocol can be obtained from Murdoch Children's Research Institute. Prior to access to any data the following would be required: a data access agreement must be signed by all relevant parties, the investigators of the study must see and approve the analysis plan describing how the data will be analysed. There must be also an agreement around appropriate acknowledgement in any future publications.
Access Criteria: The data may be obtained from the Melbourne Children's Trials Centre (MCTC) at Murdoch Children's Research Institute by emailing MCTC@mcri.edu.au.

REFERENCES:
- [Derived] Conyers R, Halman A, Moore C, Stenta T, Felmingham B, Collier L, Khatri D, Spelman T, Williams E, Dyas R, Kotecha RS, Jessop S, Mateos MK, Swen J, Elliott DA. Minimising Adverse Drug Reactions and Verifying Economic Legitimacy-Pharmacogenomics Implementation in Children (MARVEL- PIC): protocol for a national randomised controlled trial of pharmacogenomics implementation. BMJ Open. 2024 May 16;14(5):e085115. doi: 10.1136/bmjopen-2024-085115. PMID 38760050